CLINICAL TRIAL: NCT05361941
Title: Multicenter Trial of Antibiotic Eluting Graft for Promoting New Bone Growth In/near Infected Bone Cavities
Acronym: MAGIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TP-001-21
Record Dates: First submitted 2022-04-12; First posted 2022-05-05 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Periprosthetic Joint Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment Arm (Experimental): The device will be placed in voids at Stage 1. This will be followed by IV therapy for about six weeks, followed by assessment of infection, with a stage 2 surgery to follow. (For 1.5-stage, stage 2 procedure is optional). During the stage 2 surgery, the surgeon completes the procedure with affixing the revision implants.
  Interventions: Device: EP Granules with Tobramycin
- Control Arm (Active Comparator): In the standard of care arm, voids are left empty and a bone cement spacer placed during stage 1 surgery. This is followed by IV therapy for a minimum of six weeks, followed by a pathology assessment of infection by needle aspiration, after week 8, with a stage 2 surgery scheduled after week 9. During the stage 2 surgery, the spacer is removed and procedure completed by affixing the revision implants. For 1.5-stage procedures, the stage 2 procedure is optional.
  Interventions: Device: empty voids

INTERVENTIONS:
Device: EP Granules with Tobramycin — EP Granules with Tobramycin is a Ca-salt resorbable intended for orthopedic applications as a bone void filler for bone gaps or voids and in cases where risk of post-operative infection is high, such as the first stage of a 2-stage or 1.5 stage revision of an infected total joint.
  Arms: Treatment Arm
Device: empty voids — Voids are left empty
  Arms: Control Arm

SUMMARY:
This is a pivotal, prospective, multi-center, randomized, concurrent control, patient and assessor-blinded study with two arms: a treatment arm (where subjects will be treated with the EP Granules with Tobramycin investigational device in the 1st stage of a staged revision for periprosthetic joint infection (PJIs), and a control arm (where subjects are treated with the standard-of-care revision for infected PJIs).

DETAILED DESCRIPTION:
This is a pivotal, prospective, multi-center, randomized, concurrent control, patient and assessor-blinded study to demonstrate superiority of new bone growth and a reduction in recurring infections, and thereby improve outcomes for patients undergoing a staged revision for periprosthetic joint infections (PJIs).

The standard of care for treatment of PJIs typically involves either a 2-stage revision or 1.5 stage revision which entails loss of bone stock resulting from debridement of infected bone in Stage 1. In the Stage 2 procedure, surgeons use metal cones to make up for this bone loss and better support the revision implant. Inadequate bone growth could result in gaps at the the voids below the level of the cortical bone, resulting in regions with no contact with the revision implant or cement mantle. Such gaps could result in dead-space regions, and zones without new bone growth required to support the revision implant. Both deficiencies affect long-term survival of the revision implant.

The study has two arms: a treatment arm (where subjects will be treated with the EP Granules with Tobramycin investigational device in the 1st stage of the staged surgical treatment, and a control arm where subjects are treated with the standard-of-care staged surgical treatment for infected PJIs.

Outcomes are demonstration of new bone growth and reduction of recurrent infections.

ELIGIBILITY:
Inclusion Criteria:

* Ages and sexes eligible: at least 22 years, male and female
* Candidates with known infected TKA
* Life expectancy of at least 1 year
* Patient is willing to provide informed consent, is geographically stable and able to comply with the required follow up visits, testing schedule and medication regimen
* Adequate soft tissue coverage
* Signed institutional review board approved informed consent

Exclusion Criteria:

* Severe renal impairment with eGFR <50 ml/min/1.73 m2, or being treated with dialysis

  * Known hypersensitivity to aminoglycoside antibiotics, or calcium hydroxyapatite
  * Pre-existing calcium metabolism disorder
  * Uncontrolled diabetes mellitus (hemoglobin A1c levels > 8)
  * A current endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, hyperthyroid parathyroid hormone disorder, Ehler- Danlos syndrome, osteogenesis imperfecta)
  * Neuromuscular disorders such as myasthenia gravis
  * Untreated malignant neoplasm(s), or currently undergoing radiation chemotherapy
  * Inadequate neurovascular status in the involved limb that may jeopardize healing
  * HIV
  * Pregnancy
  * Adult patients requiring a legal guardian to sign informed consent form

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
A single composite outcome of new bone growth and reduction in infection rates, with absence of serious device related adverse events. | 24 months after stage 1 surgery
  A] New bone growth observed in voids at 12 months versus pre-op stage 1 and B] Absence of infection at 24 months versus pre-op stage 1 surgery.
Absence of serious device related adverse events requiring re- operation | 24 months after stage 1 surgery
  A serious device related adverse event requiring re-operation
  * Success = no adverse event occurs
  * Failure = adverse event occurs

SECONDARY OUTCOMES:
Secondary outcome: patient reported quality of life. | 12 months after stage 1 surgery
  SF-12 or PROMIS -10 score
Secondary outcome: AKSS Score | 12 months after stage 1 surgery
  1. AKSS Pain and Function Scores

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Evans, MD, Study Chair — Holy Cross Jordan Valley Hospital
Locations (12):
- United States (12):
  - University of Southern California, Los Angeles, California
  - Endeavor Health Skokie Hospital, Skokie, Illinois
  - OrthoIndy, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Womens Hospital, Boston, Massachusetts
  - U Michigan Medical Center, Ann Arbor, Michigan
  - Hospital for Special Surgery, New York, New York
  - Sanford South University Medical Center, Fargo, North Dakota
  - JIS Orthopedics, Columbus, Ohio
  - UT Health San Antonio, San Antonio, Texas
  - Jordan Valley Medical Center, West Jordan, Utah
  - West Virginia University Medical Center, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No